CLINICAL TRIAL: NCT06154421
Title: Metacarpophalangeal Joint Prostheses in Hand Surgery. A Retrospective Investigation on Functional Outcome After Intervention.
Brief Title: Metacarpophalangeal Joint Prostheses in Hand Surgery.
Acronym: FLEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Waldfriede Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BB163-23
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis Metacarpophalangeal Joint; Rheumatoid Arthritis Metacarpophalangeal Joint
Keywords: metacarpophalangeal joint prostheses; Swanson flexible finger joint implant; finger joint replacement; Osteoarthritis; Rheumatoid Arthritis; metacarpophalangeal joint arthroplasty; KeriFlex® finger joint prostheses
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis finger joint destruction: Patients with rheumatoid arthritis who received a metacarpophalangeal joint prostheses system after 01.01.2014
  Interventions: Procedure: Metacarpophalangeal joint prostheses
- Osteoarthritis finger joint destruction: Patients with post-traumatic wrist osteoarthritis who received a metacarpophalangeal joint prostheses system after 01.01.2014
  Interventions: Procedure: Metacarpophalangeal joint prostheses

INTERVENTIONS:
Procedure: Metacarpophalangeal joint prostheses — Observation after implantation of metacarpophalangeal joint prostheses using KeriFlex® or Swanson finger joint implants
  Groups: Rheumatoid Arthritis finger joint destruction
Procedure: Metacarpophalangeal joint prostheses — Observation after implantation of metacarpophalangeal joint prostheses using KeriFlex® or Swanson finger joint implants
  Groups: Osteoarthritis finger joint destruction

SUMMARY:
The primary working hypothesis of this study is whether KeriFlex® metacarpophalangeal joint prostheses provide an equivalent result to Swanson finger joint implants in patients with rheumatoid arthritis or post-traumatic osteoarthritis. Functional status will be measured by Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire no earlier than 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Metacarpophalangeal Joint Prostheses between 2014 and 2022 using Swanson or KeriFlex implant system at Hospital Waldfriede

  * rheumatoid Arthritis or post-traumatic osteoarthritis of Metacarpophalangeal joint

Exclusion Criteria:

* post surgery bone fracture of the same limb
* Pregnancy, lactation
* active malignant tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have either suffered Metacarpophalangeal joint destruction due to rheumatiod arthritis inflammation, or individuals who have received joint implant due to post-traumatic osteoarthritis of the Metacarpophalangeal joint.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand questionnaire (DASH) | All patients who underwent surgery between 2014 to 2023
  Disabilities as measured by the DASH scale; No Difficulty (1), Mild Difficulty (2), Moderate Difficulty (3), Severe Difficulty (4), Unable (5)

SECONDARY OUTCOMES:
Functional assessment: Goniometry | All patients who underwent surgery between 2014 to 2023
  ROM of each joint of the hand with a goniometer
Short-Form 36 (SF-36) | All patients who underwent surgery between 2014 to 2023
  Scored review of health questionnaire SF36: minimum value = 0 ; maximum value = 100
Ultrasound Assessment | All patients who underwent surgery between 2014 to 2023
  Patients will undergo an ultrasound scan to assess the severity of their rheumatoid arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lautenbach, MD, Study Chair — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin; Markus Bock, MD, Principal Investigator — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin
Locations (1):
- Waldfriede Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided